CLINICAL TRIAL: NCT06213116
Title: Comparing the Efficacy Between Lignocaine Given Via MADgic Atomizer and Lignocaine Pump Spray Pre Endotracheal Intubation in Adult Undergoing General Anesthesia.
Brief Title: Comparing the Efficacy Between Lignocaine Given Via MADgic Atomizer and Lignocaine Pump Spray
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Rhendra Hardy Mohamad Zaini, Asssociate Proffessor, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USM/JEPeM/21080580
Record Dates: First submitted 2023-09-27; First posted 2024-01-19 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Sore Throat; Cough; Hoarseness; Hemodynamic Instability
Keywords: lignocaine; MADgic Atomizer; airway anesthesia
MeSH Terms: conditions — Pharyngitis; Cough; Hoarseness

STUDY DESIGN:
Intervention Model Description: Prospective, randomized control study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant and Outcome Assessor do not know type of intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MADgic Atomizer (Experimental): Group M(MADgic) acting as Intervention Group:
  Patients receiving Lignocaine 30mg (3 alliquotes) given via MADgic Laryngotracheal Atomization Device prior to endotracheal intubation.
  Interventions: Device: MADgic Atomizer
- Lignocaine Spray (Active Comparator): Group S (Spray) acting as Control Group:
  Patients receiving Lignocaine 30 mg (3 puffs) given via 10mg Lignocain Pump Spray prior to endotracheal intubation.
  Interventions: Device: Lignocaine pump spray

INTERVENTIONS:
Device: MADgic Atomizer — Device to deliver directly lignocaine
  Arms: MADgic Atomizer
Device: Lignocaine pump spray — Lignocaine 30 mg (3 puffs) given via 10mg Lignocaine Pump Spray prior to endotracheal intubation
  Arms: Lignocaine Spray

SUMMARY:
Comparing the efficacy between Lignocaine given via MADgic Atomizer and Lignocaine Pump Spray pre endotracheal intubation in adult undergoing General Anesthesia.

DETAILED DESCRIPTION:
Comparing the efficacy of Lignocaine given via 2 device (Lignocaine Spray and MADGIC Atomizer) on hemodinamic parameters postintubations and severity grading of post operative sore throat, cough and hoarseness of voice.

ELIGIBILITY:
Inclusion Criteria:

* Adult with the age of 18 to 65 years old
* Gender of both male and female
* Planned for elective surgery scheduled at General Operation Theatre that require elective intubation for general anesthesia
* American Society Anaesthesiologist (ASA) preoperative physical status assessment of 1 and 2
* Airway assessment Malampati scoring 1and 2.

Exclusion Criteria:

* Pregnancy
* Known allergy or hypersensitivity to Lignocaine
* Pre existing sore throat or hoarseness of voice identified during preoperative assessment.
* The use of airway device other than endotracheal tube (ETT) such Laryngeal Mask airway/Supraglottic Device'
* Oral and neck surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Severity Grading of Post Operative Sore Throat | 24 hours
  Numbers of participants complaining incidence of sore throat postoperatively

SECONDARY OUTCOMES:
Severity Grading of Post Operative Cough | 24 hours
  Numbers of participants complaining incidence of cough postoperatively
Severity grading of Hoarseness of voice | 24 hours
  Numbers of participants complaining incidence of hoarseness of voice postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: rhendra hardy Mohamad Zaini, MD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- University of Science Malaysia Hospital, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No